CLINICAL TRIAL: NCT01759290
Title: ABSORB FIRST Registry: An International Post-market Registry of Patients With de Novo Lesions in Previously Untreated Vessels Treated With Absorb Bioresorbable Vascular Scaffold (Absorb BVS).
Brief Title: ABSORB FIRST is a Registry Designed to Evaluate the Safety and Performance of Absorb Bioresorbable Vascular Scaffold (Absorb BVS) Used in Real-world Patients.
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-302
Record Dates: First submitted 2012-12-14; First posted 2013-01-03 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Total Occlusion of Coronary Artery; Coronary Occlusion; Coronary Artery Disease; Coronary Artery Restenosis; Coronary Artery Stenosis; Coronary Disease; Coronary Restenosis
Keywords: Angioplasty; Bioabsorbable; Bioresorbable; BVS; Coronary Artery Endothelial Responsiveness; Coronary Scaffold; Coronary Stent
MeSH Terms: conditions — Coronary Occlusion; Coronary Artery Disease; Coronary Restenosis; Coronary Stenosis; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Absorb Bioresorbable Vascular Scaffold: Subjects receiving the Absorb Bioresorbable Vascular Scaffold
  Interventions: Device: Absorb Bioresorbable Vascular Scaffold

INTERVENTIONS:
Device: Absorb Bioresorbable Vascular Scaffold — Subjects receiving the Absorb Bioresorbable Vascular Scaffold

SUMMARY:
ABSORB FIRST is a prospective, multi-center registry. The objectives of the study are to:

* Provide ongoing post-market surveillance for documentation of safety, performance and clinical outcomes of the Absorb BVS (Bioresorbable Vascular Scaffold) System in daily percutaneous coronary intervention (PCI) practice per Instructions for Use (IFU, on-label use).
* To evaluate the safety and performance of 12 mm or shorter Absorb BVS in single or overlapping use (bailout, optimization of long lesion treatment) for the treatment of patients with ischemic heart disease caused by de novo native coronary artery lesion(s)
* Collect additional information (e.g. acute success) to evaluate handling and implantation of Absorb BVS by physicians under a wide range of commercial use conditions and following routine clinical practice.

DETAILED DESCRIPTION:
the ABSORB FIRST Registry is intended to provide an assessment of the safety and performance of the Absorb BVS device in accordance to the IFU in real world use involving more complex patients, lesions and use (examples: longer lesions, overlapping use, bailout, patients at high risks for cardiac events, etc.).

The ABSORB FIRST study will register a minimum of 1800 patients in approximately 90 sites throughout multiple countries worldwide where Absorb BVS has regulatory approval or is commercially available.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria must follow the most recent IFU which may include but are not limited to the following:

  * Patient must be at least 18 years of age at the time of signing the Informed Consent Form
  * Patient is to be treated for de novo lesions located in previously untreated vessels.
  * Patient must agree to undergo all required follow-up visits and data collection.

Exclusion Criteria:

* The exclusion criteria must follow the most recent IFU which may include but are not limited to the following:

  * Inability to obtain a signed informed consent from potential patient.
  * Patient belongs to a vulnerable population (per investigator's judgment, this also includes people with a direct link (hierarchical or financial benefit) to the registry Doctor or the registry Sponsor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled into this registry will be male and female patients derived from the general interventional cardiology population who satisfy the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2013-01; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Seth, MD, Principal Investigator — Fortis Escorts Heart Institute, New Delhi; Eric Eeckhout, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois; Peter Staehr, MD, Study Director — Abbott Medical Devices; Vivian Mao, MD, MPH, Study Director — Clinical Science
Locations (1):
- Abbott Vascular International BVBA, Brussels, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1800 subjects were enrolled at 87 outside US (OUS) study sites across 21 counties worldwide. The first patient registered on January 21, 2013. The patient registration was complete on Aug 30, 2014, and the last patient completed the 1-year clinical follow-up on Sep 09, 2015. The database has been closed on Oct 30, 2015.
Pre-assignment Details: A total of 81 subjects are discontinued from the study population (1800) due to death:17, withdrawal of consent:5, withdrawn by physician:2, loss to follow-up:53 and unknown reasons:4. A total of 28 subjects with MI/revascularization events or reached 1-year follow-up window were included in the clinical outcome analysis.
Period: Overall Study
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Started | 1800
Completed | 1719
Not Completed | 81
Not completed — Subjects withdrawn consent | 5
Not completed — Physician Decision | 2
Not completed — Death | 17
Not completed — Lost to Follow-up | 53
Not completed — Unknown reason | 4

BASELINE CHARACTERISTICS:
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1800
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 362
  Male | 1438
Region of Enrollment [Number; unit: participants]
  Germany | 378
  Spain | 308
  Netherlands | 144
  Belgium | 119
  Singapore | 93
  Malaysia | 88
  Thailand | 75
  Colombia | 74
  United Arab Emirates | 65
  Indonesia | 64
  France | 59
  Switzerland | 59
  Austria | 51
  New Zealand | 42
  Saudi Arabia | 39
  Jordan | 37
  Bahrain | 33
  Vietnam | 33
  Poland | 22
  Italy | 12
  Philippines | 5

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Death/TV-MI/ID-TLR (Target Lesion Failure (TLF))
Description: Target Lesion Failure includes Cardiac Death,Target Vessel-Myocardial Infarction and Ischemic Driven-Target Lesion Revascularization. This is one of the Composite Clinical Endpoints (Safety and Efficacy, hierarchical).
Time Frame: 0 to 407 days
Population: Subjects are only counted once for each type of event in each time period.The denominators used in the calculations determined according to the analysis population with excluding subjects who are lost to follow-up through given timepoint without any DMR event (all death, all MI per Protocol definition, all revascularization, respectively).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 2.8 [2.11 to 3.72]

2. Secondary Outcome: Acute Success: Clinical Device Success (Lesion Level Analysis)
Description: Device success was defined as the achievement of a final in-scaffold residual diameter stenosis of <50% assessed by online quantitative angiography or visual estimation, using Absorb BVS and without a device deficiency. A device was considered to have failed if it did not meet the requirements of the definition for clinical device success.
Time Frame: < or = 1 day
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Target Lesions
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1800
Number analyzed (Target Lesions) | 2183
percentage of lesions | 98.0 [97.30 to 98.53]

3. Secondary Outcome: Acute Success: Clinical Procedure Success (Per Subject Analysis)
Description: Procedure success was defined as the achievement of a final in-scaffold diameter stenosis of <50% by online quantitative coronary angiography (QCA) or visual estimation using Absorb BVS, with or without any adjunctive devices, and without the occurrence of cardiac death, target vessel MI (Q-wave and non-Q-wave MI), or repeat revascularization of the target lesion within 3 days of the index procedure.
Time Frame: During the hospital stay with a maximum of 3 days post index procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1800
percentage of participants | 97.0 [96.10 to 97.74]

4. Secondary Outcome: Acute Scaffold Thrombosis
Time Frame: <1 day
Population: Analysis population excludes subjects who are truly lost-to-follow-up, defined as subjects who are terminated through a given time point without any Scaffold Thrombosis event.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1770
percentage of participants
  Definite | 0
  Probable | 1
  Definite/Probable | 1

5. Secondary Outcome: Subacute ScaffoldThrombosis
Time Frame: 1 to 30 days
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1770
percentage of participants
  Definite | 9
  Probable | 2
  Definite/Probable | 11

6. Secondary Outcome: Late Scaffold Thrombosis
Time Frame: 31 to 365 Days
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1756
percentage of participants
  Definite | 5
  Probable | 2
  Definite/Probable | 7

7. Secondary Outcome: All Death, All MI, All Revascularization (DMR)
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 1.9 [1.33 to 2.67]

8. Secondary Outcome: Cardiac Death/All MI/ID-TVR (Target Vessel Failure (TVF)
Description: Target Vessel Failure (TVF) includes Cardiac Death, All Myocardial Infarction and Ischemic Driven-Target Vessel Revascularization. This is one of the Composite Clinical Endpoints (Safety and Efficacy, hierarchical).
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 1.0 [0.56 to 1.53]

9. Secondary Outcome: Major Adverse Cardiac Event (MACE)
Description: MACE includes Cardiac Death, All Myocardial Infarction and Ischemic Driven-Target Lesion Revascularization. This is one of the Composite Clinical Endpoints (Safety and Efficacy, hierarchical).
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.9 [0.52 to 1.46]

10. Secondary Outcome: Cardiac Death/TV-MI/ID-TLR (Target Lesion Failure (TLF))
Description: as for outcome 1
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.8 [0.43 to 1.32]

11. Secondary Outcome: Cardiac Death/All MI
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.8 [0.43 to 1.32]

12. Secondary Outcome: All Death/All MI
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.8 [0.43 to 1.32]

13. Secondary Outcome: All Death, All MI, All Revascularization (DMR)
Time Frame: 0 to 37 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 3.0 [2.30 to 3.96]

14. Secondary Outcome: Cardiac Death/All MI/ID-TVR (Target Vessel Failure (TVF)
Description: as for outcome 8
Time Frame: 0 to 37 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 1.4 [0.87 to 2.01]

15. Secondary Outcome: Major Adverse Cardiac Event (MACE)
Description: as for outcome 9
Time Frame: 0 - 37 Days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 1.2 [0.78 to 1.87]

16. Secondary Outcome: Cardiac Death/TV-MI/ID-TLR (Target Lesion Failure (TLF))
Description: as for outcome 1
Time Frame: 0 to 37 Days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 1.1 [0.65 to 1.67]

17. Secondary Outcome: Cardiac Death/All MI
Time Frame: 0 to 37 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 1.1 [0.69 to 1.74]

18. Secondary Outcome: All Death/All MI
Time Frame: 0 to 37 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 1.1 [0.69 to 1.74]

19. Secondary Outcome: All Death, All MI, All Revascularization (DMR)
Time Frame: 0 to 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 6.5 [5.40 to 7.76]

20. Secondary Outcome: Cardiac Death/All MI/ID-TVR (Target Vessel Failure (TVF)
Description: as for outcome 8
Time Frame: 0 to 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 2.8 [2.06 to 3.65]

21. Secondary Outcome: Major Adverse Cardiac Event (MACE)
Description: as for outcome 9
Time Frame: 0 to 180 Days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 2.4 [1.77 to 3.26]

22. Secondary Outcome: Cardiac Death/TV-MI/ID-TLR (Target Lesion Failure (TLF))
Description: as for outcome 1
Time Frame: 0 to 180 Days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 2.1 [1.53 to 2.94]

23. Secondary Outcome: Cardiac Death/All MI
Time Frame: 0 to 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 1.9 [1.29 to 2.61]

24. Secondary Outcome: All Death/All MI
Time Frame: 0 to 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 2.0 [1.43 to 2.81]

25. Secondary Outcome: All Death, All MI, All Revascularization (DMR)
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 8.4 [7.14 to 9.78]

26. Secondary Outcome: Cardiac Death/All MI/ID-TVR (Target Vessel Failure (TVF)
Description: as for outcome 8
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 3.7 [2.86 to 4.67]

27. Secondary Outcome: Major Adverse Cardiac Event (MACE)
Description: as for outcome 9
Time Frame: 0 to 407 Days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 3.1 [2.36 to 4.04]

28. Secondary Outcome: Cardiac Death/All MI
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 2.1 [1.48 to 2.88]

29. Secondary Outcome: All Death/All MI
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 2.3 [1.67 to 3.14]

30. Secondary Outcome: Death (Cardiovascular, Non-Cardiovascular)
Description: This is one of the Safety Component (non-hierarchical) endpoints.
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.1 [0.01 to 0.41]

31. Secondary Outcome: All Myocardial Infarction (MI): Q-wave MI (QMI) and Non-QMI (NQMI), TV, and Non-TV (NTV).
Description: This is one of the Safety Component (non-hierarchical) endpoints.
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.7 [0.35 to 1.18]

32. Secondary Outcome: Target Lesion Revascularization (TLR): All TLR
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.4 [0.16 to 0.81]

33. Secondary Outcome: Target Lesion Revascularization : Ischemia-Driven (ID-TLR)
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.4 [0.16 to 0.81]

34. Secondary Outcome: Target Vessel Revascularization (TVR): All TVR
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.5 [0.20 to 0.89]

35. Secondary Outcome: Target Vessel Revascularization : Ischemic-driven (ID-TVR)
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.5 [0.20 to 0.89]

36. Secondary Outcome: All Revascularization
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 7 days (In-hospital)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 1.4 [0.92 to 2.08]

37. Secondary Outcome: Death (Cardiovascular, Non-Cardiovascular)
Description: This is one of the Safety Component (non-hierarchical) endpoints.
Time Frame: 0 to 37 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.1 [0.01 to 0.41]

38. Secondary Outcome: All Myocardial Infarction (MI): Q-wave MI (QMI) and Non-QMI (NQMI), TV, and Non-TV (NTV).
Description: This is one of the Safety Component (non-hierarchical) endpoints.
Time Frame: 0 to 37 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 1.0 [0.60 to 1.60]

39. Secondary Outcome: Target Lesion Revascularization (TLR): All TLR
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 37 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.6 [0.31 to 1.11]

40. Secondary Outcome: Target Lesion Revascularization : Ischemia-Driven (ID-TLR)
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 37 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.6 [0.31 to 1.11]

41. Secondary Outcome: Target Vessel Revascularization (TVR): All TVR
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 37 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.8 [0.47 to 1.39]

42. Secondary Outcome: Target Vessel Revascularization : Ischemic-driven (ID-TVR)
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 37 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 0.8 [0.43 to 1.32]

43. Secondary Outcome: All Revascularization
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 37 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1771
percentage of participants | 2.5 [1.86 to 3.39]

44. Secondary Outcome: Death (Cardiovascular, Non-Cardiovascular)
Description: This is one of the Safety Component (non-hierarchical) endpoints.
Time Frame: 0 to 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 0.7 [0.39 to 1.25]

45. Secondary Outcome: All Myocardial Infarction (MI): Q-wave MI (QMI) and Non-QMI (NQMI), TV, and Non-TV (NTV).
Description: This is one of the Safety Component (non-hierarchical) endpoints.
Time Frame: 0 to 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 1.3 [0.83 to 1.95]

46. Secondary Outcome: Target Lesion Revascularization (TLR): All TLR
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 1.3 [0.83 to 1.95]

47. Secondary Outcome: Target Lesion Revascularization : Ischemia-Driven (ID-TLR)
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 1.3 [0.83 to 1.95]

48. Secondary Outcome: Target Vessel Revascularization (TVR): All TVR
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 1.9 [1.34 to 2.68]

49. Secondary Outcome: Target Vessel Revascularization : Ischemic-driven (ID-TVR)
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 1.8 [1.19 to 2.48]

50. Secondary Outcome: All Revascularization
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1768
percentage of participants | 5.5 [4.47 to 6.65]

51. Secondary Outcome: Death (Cardiovascular, Non-Cardiovascular)
Description: This is one of the Safety Component (non-hierarchical) endpoints.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 1.0 [0.56 to 1.54]

52. Secondary Outcome: All Myocardial Infarction (MI): Q-wave MI (QMI) and Non-QMI (NQMI), TV, and Non-TV (NTV).
Description: This is one of the Safety Component (non-hierarchical) endpoints.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 1.4 [0.92 to 2.09]

53. Secondary Outcome: Target Lesion Revascularization (TLR): All TLR
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 2.0 [1.43 to 2.81]

54. Secondary Outcome: Target Lesion Revascularization : Ischemia-Driven (ID-TLR)
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 1.9 [1.29 to 2.62]

55. Secondary Outcome: Target Vessel Revascularization (TVR): All TVR
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 2.9 [2.21 to 3.85]

56. Secondary Outcome: Target Vessel Revascularization : Ischemic-driven (ID-TVR)
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 2.6 [1.87 to 3.40]

57. Secondary Outcome: All Revascularization
Description: This is one of the Efficacy Component (non-hierarchical) endpoints.
Time Frame: 0 to 407 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Number analyzed (Participants) | 1764
percentage of participants | 7.3 [6.09 to 8.57]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Absorb Bioresorbable Vascular Scaffold
Serious Adverse Events (participants affected / at risk) | 249/1800
Other Adverse Events (participants affected / at risk) | 395/1800
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Absorb Bioresorbable Vascular Scaffold (N=1800)
Acute coronary syndrome (Cardiac disorders) | 7 (7)
Acute myocardial infarction (Cardiac disorders) | 22 (22)
Angina pectoris (Cardiac disorders) | 47 (52)
Angina unstable (Cardiac disorders) | 15 (15)
Aortic valve disease mixed (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 9 (9)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 6 (6)
Cardiac failure acute (Cardiac disorders) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 15 (17)
Coronary artery dissection (Cardiac disorders) | 6 (6)
Coronary artery occlusion (Cardiac disorders) | 2 (2)
Coronary artery perforation (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 20 (21)
Coronary artery thrombosis (Cardiac disorders) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (5)
Myocarditis (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 5 (5)
Pericardial haemorrhage (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Chest discomfort (General disorders) | 3 (3)
Chest pain (General disorders) | 12 (13)
Death (General disorders) | 2 (2)
Device malfunction (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 17 (18)
Sudden cardiac death (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 9 (11)
Jaundice (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Primary amyloidosis (Immune system disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative abscess (Infections and infestations) | 1 (1)
Prostatic abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 3 (3)
Renal haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Cardiac enzymes increased (Investigations) | 6 (6)
Cardiac stress test abnormal (Investigations) | 2 (2)
Electrocardiogram change (Investigations) | 2 (2)
Exercise electrocardiogram abnormal (Investigations) | 1 (1)
Stress echocardiogram abnormal (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (2)
Personality disorder (Psychiatric disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Aneurysm (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 3 (3)
Arterial stenosis (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 5 (5)
Hypertension (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 6 (6)
Ischaemia (Vascular disorders) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Absorb Bioresorbable Vascular Scaffold (N=1800)
Accelerated idioventricular rhythm (Cardiac disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 8 (10)
Acute myocardial infarction (Cardiac disorders) | 22 (22)
Angina pectoris (Cardiac disorders) | 69 (76)
Angina unstable (Cardiac disorders) | 17 (17)
Aortic valve disease mixed (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 16 (16)
Atrial flutter (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 7 (7)
Cardiac failure acute (Cardiac disorders) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 19 (21)
Coronary artery dissection (Cardiac disorders) | 10 (10)
Coronary artery occlusion (Cardiac disorders) | 5 (5)
Coronary artery perforation (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 33 (35)
Coronary artery thrombosis (Cardiac disorders) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 3 (3)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (5)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 10 (10)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 6 (6)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 3 (3)
Chest pain (General disorders) | 16 (17)
Death (General disorders) | 2 (2)
Device failure (General disorders) | 1 (1)
Device malfunction (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Feeling abnormal (General disorders) | 1 (1)
Malaise (General disorders) | 3 (3)
Multi-organ failure (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 34 (40)
Oedema peripheral (General disorders) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 9 (11)
Jaundice (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Primary amyloidosis (Immune system disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative abscess (Infections and infestations) | 1 (1)
Prostatic abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 3 (3)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Renal haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Cardiac enzymes increased (Investigations) | 69 (69)
Cardiac stress test abnormal (Investigations) | 2 (2)
Electrocardiogram change (Investigations) | 3 (3)
Exercise electrocardiogram abnormal (Investigations) | 3 (3)
Stress echocardiogram abnormal (Investigations) | 1 (1)
Troponin I increased (Investigations) | 8 (8)
Troponin T increased (Investigations) | 1 (1)
Troponin increased (Investigations) | 14 (14)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebellar embolism (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 7 (7)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (2)
Panic attack (Psychiatric disorders) | 1 (1)
Personality disorder (Psychiatric disorders) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (19)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hospitalisation (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 3 (3)
Arterial stenosis (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 5 (5)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Hypertensive crisis (Vascular disorders) | 6 (6)
Ischaemia (Vascular disorders) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days